CLINICAL TRIAL: NCT06361901
Title: Comparison of Therapeutic Effect and Brain Activity According to Language Rehabilitation Program and Language Therapy in Patients With Speech Impairment After Stroke. Prospective, Randomized, Single-blind, Exploratory Clinical Study
Brief Title: Comparison of Therapeutic Effect Between Speech Rehabilitation Program and Speech Therapy in Stroke Patients With Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Yang, Seung Nam, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023GR0452
Record Dates: First submitted 2023-11-27; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Aphasia; Speech Therapy
MeSH Terms: conditions — Stroke; Aphasia; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Language therapy group with language rehabilitation program (Experimental): In addition to 5-session conventional language therapy, we provide a 5-session language rehabilitation program using an AI-based computerized cognitive and language training program. A cognitive evaluation is conducted before starting treatment, and K-Western Aphasia Battery and Functional Near infrared spectroscopy are performed before and after the treatment.
  Interventions: Device: Zenicog;language rehabilitation program; Procedure: Conventional language rehabilitation
- Conventional language therapy group (Active Comparator): We provide a 10-session conventional language therapy. A cognitive evaluation is conducted before starting treatment, and K-Western Aphasia Battery and Functional Near infrared spectroscopy are performed before and after the treatment.
  Interventions: Procedure: Conventional language rehabilitation

INTERVENTIONS:
Device: Zenicog;language rehabilitation program — This program is an AI-based computerized cognitive and language training program.
  Arms: Language therapy group with language rehabilitation program
Procedure: Conventional language rehabilitation — Conventional language rahabilitation therapy will apply for all participants with speech impairement

SUMMARY:
Our study will provide precise and intensive speech rehabilitation treatment program to patients with speech disorders after stroke, and compare clinical evaluations with the conventional speech therapy patient group.

Clinical evaluation tools will be performed before and after the treatment for all patients

* K-Western Aphasia Battery for aphasia assessment tools
* Cerebral blood flow changes with near-infrared spectroscopy

DETAILED DESCRIPTION:
During the initial evaluation of this study, the patient's gender, age, and onset of stroke lesion occurrence are collected and a cognitive evaluation is performed. In addition, the K-Western Aphasia Battery for aphasia assessment tools(K-WAB) and Cerebral blood flow changes with near-infrared spectroscopy will be performed. All participants will be assigned to a test group or control group. In addition to the existing speech rehabilitation treatment, the test group will receive a speech rehabilitation program, and the control group will receive the same treatment as the existing speech rehabilitation treatment.

After treatment is completed, the K-WAB test and near-infrared spectroscopy will be performed again.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 years old
* Those with speech disorders that occurred after a stroke was diagnosed
* Those who can follow the clinical study procedures
* Those who voluntarily signed the consent form

Exclusion Criteria:

* Patients who have difficulty to consent to research and participate in speech rehabilitation programs due to cognitive decline

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Aphasic quatient | Evaluate two times ; Before speech therapy treatment program (baseline) and within 7days after the treatment period.
  Aphasic quatient using K-Western Aphasia Battery for aphasia assessment tools

SECONDARY OUTCOMES:
Change of cerebral blood flow | Evaluate two times ; Before speech therapy treatment program (baseline) and within 7days after the treatment period.
  Change of cerebral blood flow with near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, Korea University Guro Hospital, Seoul, South Korea